CLINICAL TRIAL: NCT06749522
Title: Radiological Spectrum Of Fatty Liver Correlate With High Resolution Ultrasonography Of Fibrosis And Cirrhosis
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/038
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Fibrosis; Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: high resolution ultrasonography — to compare high resolution ultrasonography finings with other imaging modalities(CT and MRI)

SUMMARY:
Fatty liver is a condition in which fat builds up in liver. it is very common health issue.it is major public health problems in the world. there is particular concern because fatty liver causes mortality among patients. The incidence and prevalence of disease vary with time. Fibrosis is thickening of connective tissues which is usually as a result of injury and long term inflammation. Cirrhosis is severe scarring of liver which is caused by long term liver damage. The scar tissue replaces healthy tissues which leads to loss of liver function. The Objective of study is to look into radiographic features of fatty liver disease. The high resolution ultrasonography will give more detailed view of disease. The study inclued 150 participants.

DETAILED DESCRIPTION:
The other liver conditions like fibrosis and cirrhosis are also examined and correlated with fatty liver disease. The CT and MRI are used to compare with HR ultrasonographic findings. Descriptive statistics and comparative statistics are used to interpret data.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of fatty liver (steatosis), fibrosis, or cirrhosis.
* Patient consent to undergo imaging and participate in the study.

Exclusion Criteria:

* Other Liver Diseases: Exclusion of patients with other significant liver conditions (e.g., viral hepatitis, autoimmune liver diseases) unless specified.
* Pregnant women may be excluded due to imaging concerns.
* Poor quality or incomplete imaging studies.
* Presence of other severe systemic illnesses that could affect liver function or imaging.
* Recent liver surgeries or invasive procedures that might affect imaging results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: to compare the Radiological Spectrum Of Fatty Liver Correlate With High Resolution Ultrasonography (CT, MRI) Of Fibrosis And Cirrhosis
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
CT | 12 Months
  CT used for the image comparision
MRI | 12 Months
  CT used for the image comparision

CONTACTS AND LOCATIONS:
Locations (1):
- AL-NAWAZ HOSPITAL,Tillu Road, Saddiqabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No